CLINICAL TRIAL: NCT04613960
Title: Magnesium in Treating Subarachnoid Hemorrhage Related Vasospasm, A Haptoglobin Genomic Based Randomized Controlled Trial
Brief Title: Magnesium Treating Subarachnoid Hemorrhage Vasospasm
Acronym: MATSH-SHapE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Collaborators: Ain Shams University (Other); Health Insurance Organization, Egypt (Unknown)
Responsible Party: Principal Investigator, Ahmed Mohammed Ateia, Neurology Specialist, MTH; Associate member, Harvard Medical School., General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTH/NEUR/20/01
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Cerebral Vasospasm
Keywords: subarachnoid hemorrhage; Haptoglobin; Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium arm (Active Comparator): patients randomized to magnesium therapy at a fixed daily dose of 64 mmol reconstituted in 0.9% saline via continuous intravenous infusion for 14 days after hemorrhage onset, or until discharge or death if it occurred.
  Interventions: Drug: Magnesium sulfate
- Placebo arm (Placebo Comparator): patients randomized to placebo therapy with 0.9% saline (without active component) via same protocol.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Magnesium sulfate — MgSO4 (at a fixed daily dose of 64 mmol reconstituted in 0.9% saline) via continuous intravenous infusion for 14 days after onset
  Arms: Magnesium arm
Drug: normal saline — Placebo treatment
  Arms: Placebo arm

SUMMARY:
A randomized clinical trial investigating magnesium sulphate ability to reduce risk of cerebral vasospasm after acute subarachnoid hemorrhage hence improving outcome particularly in haptoglobin 2-2 patients who are highly susceptible for severe complications after subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Study Design and Location:

Investigators propose a double blinded, randomized (1:1), placebo-controlled, multicenter, clinical trial including patients with acute aSAH. Participants will be allocated either to MgSO4 or placebo. The permission to conduct the study protocol will be considered for approval by the ethics committee of General Committee of Teaching Hospitals and Institutes (GCTHI), Egypt. The study will be conducted in 3 centers; El-Materia Educational Hospital, Ain Shams University Hospitals and Nasr City Insurance Hospital. The assigned centers for this study represent large-volume referral stroke centers that provide comprehensive management protocols for aSAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* age over 18 years old
* diagnosis of acute aSAH (≤ 48 hours) confirmed with angiographic evidence of cerebral aneurysm and CT brain on admission.

Exclusion Criteria:

* subarachnoid hemorrhage due to non-aneurysmal causes
* cerebral stroke of any type during past month
* decompensated heart failure, renal failure or hepatic failure
* difficult bilateral transtemporal transcranial Doppler (TCD) insonation of intracranial arteries due to thick temporal bone of the skull.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Clinical evidence and TCD measured MFV indicative of vasospasm | 14 days after onset
  Mean flow velocity measurements by TCD indicative of cerebral vasospasm. New clinical neurological deficit determined by comparing NIHSS pre and post detected vasospasm.

SECONDARY OUTCOMES:
Poor MRS functional score | 3 months after the onset
  Poor MRS score (4,5 or dead) assessed at regular follow up visits

CONTACTS AND LOCATIONS:
Locations (1):
- El matareya Educational Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Reddy D, Fallah A, Petropoulos JA, Farrokhyar F, Macdonald RL, Jichici D. Prophylactic magnesium sulfate for aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis. Neurocrit Care. 2014 Oct;21(2):356-64. doi: 10.1007/s12028-014-9964-0. PMID 24619389
- [Background] Soliman R, Zohry G. [Effect of magnesium sulphate and milrinone on cerebral vasospasm after aneurysmal subarachnoid hemorrhage: a randomized study]. Braz J Anesthesiol. 2019 Jan-Feb;69(1):64-71. doi: 10.1016/j.bjan.2018.09.005. Epub 2018 Nov 6. PMID 30409409
- [Background] Thomsen JH, Etzerodt A, Svendsen P, Moestrup SK. The haptoglobin-CD163-heme oxygenase-1 pathway for hemoglobin scavenging. Oxid Med Cell Longev. 2013;2013:523652. doi: 10.1155/2013/523652. Epub 2013 May 27. PMID 23781295
- [Background] Milman U, Blum S, Shapira C, Aronson D, Miller-Lotan R, Anbinder Y, Alshiek J, Bennett L, Kostenko M, Landau M, Keidar S, Levy Y, Khemlin A, Radan A, Levy AP. Vitamin E supplementation reduces cardiovascular events in a subgroup of middle-aged individuals with both type 2 diabetes mellitus and the haptoglobin 2-2 genotype: a prospective double-blinded clinical trial. Arterioscler Thromb Vasc Biol. 2008 Feb;28(2):341-7. doi: 10.1161/ATVBAHA.107.153965. Epub 2007 Nov 21. PMID 18032779
- [Result] Ateia AM, Elbassiouny A, El-Nabi SH, Fahmy NA, Ibrahim MH, El-Garawani I, Geba KM, Khalaf M. Predictive value of haptoglobin genotype as a risk of cerebral vasospasm after aneurysmal subarachnoid hemorrhage. Clin Neurol Neurosurg. 2020 Dec;199:106296. doi: 10.1016/j.clineuro.2020.106296. Epub 2020 Oct 7. PMID 33069930